CLINICAL TRIAL: NCT06938633
Title: Utility of Urine Mass Spectrometry Analysis in Addressing Medication Non-adherence in Patients With Poorly Controlled Hypertension
Brief Title: Addressing Medication Non-adherence in Patients With Poorly Controlled Hypertension Using Urine Mass Spectrometry
Acronym: ADURINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADURINE
Record Dates: First submitted 2023-12-05; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-01

CONDITIONS: Hypertension; Uncontrolled Hypertension; Non-Adherence, Medication
Keywords: Urine mass spectrometry; Uncontrolled hypertension; Medication non-adherence
MeSH Terms: conditions — Hypertension; Medication Adherence | interventions — Gas Chromatography-Mass Spectrometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mass spectrometry analysis (Experimental): All patients will be collected 50mls of urine for mass spectrometry analysis to determine medication adherence during each study visit; on enrolment, at 3-month, and at 6-month period.
  Interventions: Other: mass spectrometry analysis

INTERVENTIONS:
Other: mass spectrometry analysis — The collected urine samples will be analyzed to determine medication adherence during study visits

SUMMARY:
* Hypertension is the single largest contributor to cardiovascular disease and death. While adequate control of hypertension reduces risk of disease, many patients have uncontrolled hypertension. This is often due to medication non-adherence. Left undetected, patients are prescribed additional medications, and referred to multiple specialists for investigations - leading to increased healthcare costs. Hence, detecting non-adherence to antihypertensive medications is important. However, patient history, patient recall, or questionnaires, are often inaccurate. Most recently, urine measurements of antihypertensive drug levels, using mass spectrometry, has been established as the gold standard to assess medication adherence. The one-time urine test for medication adherence is ideal: It's convenient, non-invasive, economical, and can be easily performed in a clinic setting. By improving blood pressure control, this will lead to reductions in healthcare visits, avoidance of catastrophic cardiovascular events. Ultimately, this translates to significant economic savings for both patients with hypertension and the healthcare system.
* Therefore, the investigators hypothesize that the implementation of urine adherence testing coupled with targeted counselling will improve the adherence and blood pressure control in hypertension. To do this, the investigators aim to (1) evaluate for medication adherence in 312 participants with recent stroke and hypertension; (2) evaluate for medication non-adherence in participants with uncontrolled hypertension; and (3) assess if detection of non-adherence can improve hypertension control.

DETAILED DESCRIPTION:
• The investigators plan to achieve these aims in three steps. First, the investigators retrospectively assess medication adherence in 200 participants admitted for recent stroke using urine biospecimens collected. Second, the investigators will prospectively recruit 100 participants with poorly controlled hypertension and assess for medication adherence. Finally, participants detected with non-adherence will be counselled. These participants will be reassessed for improvements in both medication adherence and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 21 - 80 years
2. Systolic blood pressure of ≥140 mmHg or average systolic blood pressure ≥135 mmHg, or diastolic blood pressure ≥90 mmHg or average diastolic blood pressure ≥85 mmHg, on at least two measurements
3. Currently taking 2 or more hypertension medications
4. Able to provide informed consent.

Exclusion Criteria:

* Significant kidney impairment with eGFR of less than 45mL/min/1.73m2 or on dialysis
* Known history of chronic liver disease

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in adherence rate | 6 months
  This is the difference in the adherence rates at enrollment and at the end of the study
The change in systolic blood pressure | 6 months
  This is the difference in systolic blood pressure between enrollment and the last follow up visit at 6 months
The change in diastolic blood pressure | 6 months
  This is the difference in diastolic blood pressure between enrollment and the last follow up visit at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No